CLINICAL TRIAL: NCT02199301
Title: Tolerance Induction in Living Donor Kidney Transplantation With Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-07-210
Record Dates: First submitted 2012-09-10; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2012-09

CONDITIONS: End Stage Renal Disease
Keywords: Kidney transplantation; Tolerance induction; Immunosuppression withdrawal; Bone marrow transplantation; Transplantation conditioning; Hematopoietic stem cell transplantation; Living donor; Haplotype; Immune tolerance
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation Conditioning

ARMS (1):
- BMTKT (Experimental): Transplantation Conditioning for bone marrow transplantation (BMT) Kidney transplantation and BMT (BMTKT)
  Interventions: Procedure: Transplantation Conditioning for BMT

INTERVENTIONS:
Procedure: Transplantation Conditioning for BMT — Transplantation Conditioning for BMT (POD#-7~-1) POD#-7: Rituximab (Mabthera, Roche Pharma Aktiengesellschaft (AG) Swiss) 375/m2 iv infusion POD#-6~-3: Fludarabine (Fludara Inj., Bayer AG, Germany) 30mg/m2/day iv infusion POD#-5~-4: Cyclophosphamide (Endoxan Inj., Baxter Oncology Gesellschaft mit beschränkter Haftung (GmbH), Germany) 30mg/kg/day iv infusion POD#-2: (Rituximab 375/m2 iv infusion) POD#-1: Thymic irradiation (Dose, 700cGy)

SUMMARY:
Kidney transplantation (KT) requires a life-long immune suppression (IS). It has been well-known that long-term IS inevitably causes various complication e.g. infection, toxicity, diabetes, osteoporosis, avascular necrosis of hip joint, cataract, acne, and malignancies and so on. Tolerance induction showing graft function without maintenance IS has been considered as a final solution in the transplantation recipients. Tolerance induction can be achieved in KT recipients with donor hematopoietic stem cell transplantation (HSCT).

In this study, adult patients (18 and more years of age) with a human leukocyte antigen (HLA)-haplotype match donor are enrolled. Patients receive preconditioning treatment for HSCT 1week prior to KT. Bone marrow is harvested from donor under general anesthesia at the time of nephrectomy for transplantation in donor. Donor BM is infused immediate post-transplantation at intensive care unit (ICU). Immunologic measurements including microchimerism study and protocol biopsy will be followed at several time points. IS will be tapered slowly and withdrawn over a period of several months.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adult (18 and more years of age) living donor kidney transplant recipients who have a one haplotype match donor.
2. Patients who have no known contraindication to administration of rabbit anti-thymocyte globulin (ATG) or radiation.
3. Patients who agree to participate in the study and sign an Informed Consent.

Exclusion Criteria:

1. Presence of previous episode of transplantation including kidney
2. Simultaneous multi-visceral transplantation
3. Demonstration of donor specific antibody (DSA) or panel reactive antibody(PRA) greater than 20%
4. ABO blood type incompatible
5. Previous treatment with rabbit anti-thymocyte globulin or a known allergy to rabbit proteins.
6. History of malignancy with the exception of non-melanoma skin malignancies.
7. Uncontrolled systemic or concomitant unstable infection
8. Serological evidence of Hepatitis B or Hepatitis C or HIV infection.
9. Severe psychiatric disease
10. Leukopenia (with a white blood cell count < 3000/mm3)
11. Disagreement to participate in the study and sign an Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Immune Suppression Withdrawal | Immune Suppression Withdrawal within 18 months post-transplantation
  Immune suppression will be tapered-off and withdrawn over the period of 6 to 18 months post-transplantation under the monitoring of graft function and immunologic measurements.

SECONDARY OUTCOMES:
Graft failure | At the post-transplantation 18 months
  In this study, immune suppression(IS) will be tapered-off and withdrawn over the period of 6 to 18 months post-transplantation under the monitoring of graft function and immunologic measurements. At the post-transplantation 18 months we evaluate graft failure episode irrespective of IS withdrawal.
Allograft Rejection | At the post-transplantation 18 months
  In this study, immune suppression(IS) will be tapered-off and withdrawn over the period of 6 to 18 months post-transplantation under the monitoring of graft function and immunologic measurements. At the post-transplantation 18 months we evaluate allograft rejection episode irrespective of IS withdrawal.

OTHER OUTCOMES:
Microchimerism | At post-transplantation 1, 2, 3, 4, 8, and 24 wks
  Presence and proportion of microchimerism in recipient's peripheral blood will be measured by microsatellite short tandem repeat.
Immune Cell Profiling | At post-transplantation 1, 2, 4, 8, 12, 24, and 52 weeks
  Changes of proportion or absolute count of immune cells are measured by flowcytometric analysis in recipient's peripheral blood, using cluster of differentiation (CD) marker.
Mixed Lymphocyte Reaction | At post-transplantation 8, 24, 52 weeks
  Mixed lymphocyte reaction will be done for the evaluation for the donor-specific immune response (Donor vs. 3rd party) in vitro.
Protocol Biopsy | Post-transplantation 3, 24, and 52 weeks
  Absence or presence of allograft rejection is confirmed by ultrasonography-guided percutaneous biopsy during follow-up and prior to withdrawal of immunosuppressive agent.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Organ Transplant Center, Seoul, South Korea